CLINICAL TRIAL: NCT04118894
Title: Wright Foot & Ankle Post-Market Observational Study
Status: Terminated | Type: Observational
Why Stopped: Due to COVID the enrollment into the study was delayed. Sponsor chose to collect clinical data via alternative methods.
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: INT19-MDR-001
Record Dates: First submitted 2019-08-21; First posted 2019-10-08 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Arthritis; Rheumatoid Arthritis; Fracture; Trauma Injury; Fusion of Joint
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Fractures, Bone; Accidental Injuries; Ankylosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Foot and Ankle Devices: The study subjects included are those treated with one or more approved or cleared Wright Medical products included in this study.
  Interventions: Device: Foot and Ankle Devices

INTERVENTIONS:
Device: Foot and Ankle Devices — Wright devices used in foot and ankle procedures

SUMMARY:
WRIGHT FOOT & ANKLE POST-MARKET OBSERVATIONAL STUDY, Multi-Year, Multi-Site, Multi-Device, Post-Market Observational Study, 10 sites, a minimum of 40 patients per device

DETAILED DESCRIPTION:
The selected design is a global, multi-center, non-randomized, prospective observational study. The study subjects included are those treated with one or more approved or cleared Wright Medical products included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to consent to participate (written, informed consent);
* Willing and able to attend/complete the requested follow-up visits;
* Considered for treatment with one or more approved or cleared Wright Medical products included in this study

Exclusion Criteria:

* Subjects determined, by the investigator, to be an inappropriate candidate for the procedure indicated;
* Unable to consent to participate (written, informed consent);
* Unable to attend/complete the requested follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Instructions for Use (IFU) for each individual product can be found at http://www.wright.com/prescribing-use-3.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (5):
- United States (2):
  - Mercer-Bucks Orthopaedics, Hamilton, New Jersey
  - OrthoCarolina, Charlotte, North Carolina
- CHRU Tours, Hôpital Trousseau, Tours, France
- Hessingpark Clinic, Augsburg, Germany
- Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 119 subjects were enrolled and treated with a study device at 5 sites in the private clinic and hospital setting in the France, Germany, United States and United Kingdom. A subject may have received more than one of the devices under investigation. The first subject was enrolled on January 22, 2020 (aligned with protocol) and the last subject was enrolled on November 1, 2021.
Pre-assignment Details: No specific method (such as randomization, blinding or stratification) for assigning subjects was used in this protocol. Consecutive subjects at each site meeting all the eligibility criteria were enrolled in this study.
Period: Overall Study
Arm/Group | Foot and Ankle Devices
Started | 119
Completed | 84
Not Completed | 35
Not completed — Lost to Follow-up | 21
Not completed — Withdrawal by Subject | 10
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Foot and Ankle Devices
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.49 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Smoking Status [Count of Participants; unit: Participants]
  Never | 77
  Previous | 38
  Current, <= 1 Pack/day | 3
  Current, > 1 pack/day | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.18 (5.58)

OUTCOME MEASURES:

1. Primary Outcome: EuroQol (EQ-5D-5L).
Description: Comparing the changes in patient-reported pain and social interaction for quality of life from pre-op through post-operatively, assessed by the EuroQol (EQ-5D-5L).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. Health utility values generated from the EQ-5D generally range from 0 (death) to 1 (perfect health). But health utility values less than 0 are possible, and represent health states considered worse than death.
  The EQ VAS records the patient's self-rated health on a VAS (0-100), where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale- EQ5D VAS
Arm/Group | Foot and Ankle Devices
Number analyzed (Participants) | 84
units on a scale- EQ5D VAS | 74.1 (22.5)

2. Secondary Outcome: Foot and Ankle Ability Measure (FAAM)
Description: Comparing the changes in patient-reported function scores from pre-op through post-operatively, assessed by the FAAM
  The FAAM is a patient-completed instrument that consists of an "Activities of Daily Living" subscale (21 scored items) and a "Sports" subscale (7 scored items) in which the response options are presented as 5-point Likert scales (range 4 to 0). Scores for each subscale range from 0% (least function) to 100% (most function).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale- FAAM SANE
Arm/Group | Foot and Ankle Devices
Number analyzed (Participants) | 82
score on a scale- FAAM SANE | 68.6 (25.5)

3. Secondary Outcome: Safety Assessment
Description: Identifying and reporting the safety of the implant in terms of complications and adverse events. (This is reported in the Adverse Event Section)
Time Frame: 1 year
Population: Safety is reported in the adverse event section.
Measure: Count of Participants; unit: Participants
Arm/Group | Foot and Ankle Devices
Number analyzed (Participants) | 119
Participants
  Subjects that Experienced a Serious Adverse Event | 9
  Subjects that Didn't Experience a Serious Adverse Event | 110

4. Secondary Outcome: Surgeon Survey
Description: Conducting a surgeon survey including radiographic assessment of fusion and consolidation time
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Foot and Ankle Devices
Number analyzed (Participants) | 112
Participants
  Wright product performed as intended- Yes | 109
  Wright product performed as intended- No | 3

5. Secondary Outcome: Patient Survey
Description: Conducting patient surveys to assess current implant status (to include complications)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Foot and Ankle Devices
Number analyzed (Participants) | 49
Participants
  Experienced any complications associated with your procedure requiring you to seek medical care?: Yes | 7
  Experienced any complications associated with your procedure requiring you to seek medical care?: No | 42
  Any surgery to remove any device parts associated with your foot/ankle procedure?: Yes | 1
  Any surgery to remove any device parts associated with your foot/ankle procedure?: No | 48

ADVERSE EVENTS:
Time Frame: Surgery to 1 year
Description: Procedural and device related events will be described and collected on the AE form. It is the responsibility of the operating surgeon/s to be aware and note the adverse effects from the package insert/instructions for use by the manufacturer/sponsor.
Arm/Group | Foot and Ankle Devices
All-Cause Mortality (participants affected / at risk) | 0/119
Serious Adverse Events (participants affected / at risk) | 9/119
Other Adverse Events (participants affected / at risk) | 19/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foot and Ankle Devices (N=119)
acute aortic dissection (Cardiac disorders) | 1 (1)
Below Knee Amputation (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (Musculoskeletal and connective tissue disorders) | 4 (5)
Non-Union (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foot and Ankle Devices (N=119)
Pain (Musculoskeletal and connective tissue disorders) | 12 (14)
Algodystrophy (Musculoskeletal and connective tissue disorders) | 1 (1)
Blister Dorsal Aspect of Operated Foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Inflammatory Scar (Musculoskeletal and connective tissue disorders) | 1 (1)
Wound Healing Complications (Musculoskeletal and connective tissue disorders) | 5 (5)
Ulcer (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04118894/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04118894/SAP_001.pdf